CLINICAL TRIAL: NCT04991285
Title: People of Color and Dermatology: A Deeper Look at Patients' Perceptions of Care and the Need for Greater Diversity in Dermatology
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: STU00214929
Record Dates: First submitted 2021-07-21; First posted 2021-08-05 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Dermatology
Keywords: People of color, dermatology training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surveys will be collected to evaluate views from people of color and their dermatology experience. The information collected will look at patients' perceptions of care and the need for greater diversity in dermatology.

DETAILED DESCRIPTION:
This survey looks to gain a much-needed perspective from POC in order to better understand their views on 1. the field of dermatology 2. the diversity in dermatology and its acceptance of skin of color and hair 3. skin of color centers 4. Race concordant dermatology and 5. perceived views on dermatologic training. The sample size will be the number of participants that respond to the survey, with a target sample size of 1000 respondents. Eligible participants need to identify with at least one of the following groups

* Black or African American
* Latinx
* American Indian or Alaska Native
* Native Hawaiian or Pacific Islander
* Asian

Participants will need to be over the age of 18 years old, English-speaking/English proficient and anticipated to be living within the United States. Recruitment and screening will be done through ResearchMatch.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants need to identify with at least one of the following groups

* Black or African American
* Latinx
* American Indian or Alaska Native
* Native Hawaiian or Pacific Islander
* Asian
* Over the age of 18 years old
* English-speaking/ English proficient
* Anticipated to be living within the United States

Exclusion:

Subjects who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People of color who are over the age of 18 years old, English speaking/ English proficient and living in the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency (percentage) of participants with knowledge of skin of color clinics/training | 2 months
  The frequency (percentage) of participants who responded as knowing about skin of color clinics and skin of color training for dermatology.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Fienberg School of Medicine Department of Dermatology, Chicago, Illinois, United States